CLINICAL TRIAL: NCT02623283
Title: Assessing the Long-term Effects of a School-to-home Childhood Supervised Brushing Programme in Young Adults From High Caries Risk Groups - The Tayside Brushing Study Adult Follow up
Brief Title: The Tayside Brushing Study - Adult Follow up
Status: Completed | Type: Observational
Sponsor: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Dr Morag Curnow, Clinical Dental Director, NHS Tayside
Other Study IDs: 186595
Record Dates: First submitted 2015-11-19; First posted 2015-12-07 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention given — Participants will have a full dental examination but no operative intervention

SUMMARY:
Historically dental health of Scottish children had been poor for many years. Evidence form clinical trials of fluoride toothpaste identified a route to improving prevention. Those who had poor dental health used fluoride toothpaste infrequently at home. The investigators hypothesised that this disadvantage could be overcome by supplying toothpaste to disadvantaged families and supervising child toothbrushing at school. In 1997, 534 children 5.3 years were recruited in 12 primary schools in Tayside; randomly assigned to one of two groups - test group followed a home-to-school toothbrushing programme with fluoride toothpaste; control group: usual care. Children in test group were provided with toothbrushes and toothpaste (1,000ppmF as sodium monofluorophosphate) for home use; also brushed their teeth school daily. After 2 years, children participating in the supervised brushing programme developed significantly less caries (tooth decay).

Permission was given for longitudinal follow up of children and dental records. The original intervention lasted 30 months and children were re-examined at 36 months after baseline, 48, 60 and 84 months. At 84 month examination, 77% were available, found prolonged benefits of brushing programme. This was 4.5 years after the end of the programme; children were aged 11.5 years. At age 14 years, 6.5 years after intervention end, 65% of children were reexamined; benefit was still evident at 20-26% less caries experience. However, there had been greater subject loss and insufficient funds available to undertake a more individual followup of participants.

Since then, records have been followed; up-to-date contact details identified. Using this new data, the investigators seek to reconsent the participants, now aged 23 to invite them to attend a followup dental examination. This study has the potential to provide unique information on longterm costs and benefits of a home-to-school toothbrushing programme.

DETAILED DESCRIPTION:
Participants on the original trial will be sent an information letter and information leaflet and consent form in the post. The letter will provide contact details for the chief investigator (CI) should they wish to discuss the study before making a decision about whether they would like to take part. The letter will ask participants to complete the informed consent form and return it to the Chief Investigator in the pre-paid envelope provided. If participants do not respond to the first letter a second will be sent two weeks later. No further letters will be sent.

The consent form will ask participants to give details of which days and times are most convenient for them to attend an appointment (evening and weekend appointments will be offered). The letter will advise people that attendance does not replace their usual dental care visits. For those who do not have a dentist and wish to find one, appropriate advice and assistance will be provided by the CI, or a member of the Dental Team.

Participants who return their consent forms will be contacted by telephone by a member of the NHS Tayside dental team to arrange an appointment at a time convenient to them. If participants are unable to travel to the two centres (Broxden Dental Centre in Perth or Kings Cross Dental Department in Dundee) they may be offered a home visit.

When participants attend for their appointment they will be asked to confirm their consent verbally. Dr Morag Curnow (the same dentist that examined the participants when they were in School on the original toothbrushing trial) or another appropriately trained Dentist (named on the study delegation log) will conduct a short dental examination, recording the presence of plaque on anterior teeth and the caries status of each tooth surface using dental lighting and fibre-optic transillumination. The examining dentist will be unaware of which study group the adults belonged to when they were child participants in the trial. Participants will also be asked to complete oral health related questionnaires. Questionnaires will be analysed by a statistician.

Participants will be asked to give consent for their dental records to be accessed using health service records to record dental treatment history. Consent will be recorded in writing. Approval has already been provided by Information Services Division (ISD), NHS National Services Scotland to access the dental treatment records.

ELIGIBILITY:
Inclusion Criteria:

* A participant on the original Tayside Brushing Study

Exclusion Criteria:

-

Ages: 24 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults aged 25 who were enrolled on the Tayside Brushing Study Randomised Controlled Trial
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Caries experience (The number of each participant's Decayed, Missing and Filled Teeth (DMFT)) | Over an eight week period, each participant will be examined once
  The number of each participant's Decayed, Missing and Filled Teeth (DMFT), recorded by and extrapolated from surfaces (DMFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Broxden Dental Centre, Perth, Scotland, United Kingdom